CLINICAL TRIAL: NCT01868464
Title: Phase I Open-Label Dose Escalation Trial for the Development of a Human BCG Challenge Model for Assessment of TB Immunity
Brief Title: Challenge Model for Assessment of Human TB Immunity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0033
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2017-07-19

CONDITIONS: Tuberculosis
Keywords: challenge; Mycobacterium tuberculosis; parent protocol; TB; Tice BCG; tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BCG 16x10^6 CFU (Experimental): 30 subjects, one dose of Tice BCG intradermally, 16x10^6 cfu
  Interventions: Biological: BCG TICE strain
- BCG 2x10^6 CFU (Experimental): 30 subjects, one dose of Tice Bacillus Calmette-Guerin vaccine (BCG) intradermally, 2x10^6 colony forming units (cfu)
  Interventions: Biological: BCG TICE strain
- BCG 4x10^6 CFU (Experimental): 30 subjects, one dose of Tice BCG intradermally, 4x10^6 cfu
  Interventions: Biological: BCG TICE strain
- BCG 8x10^6 CFU (Experimental): 30 subjects, one dose of Tice BCG intradermally, 8x10^6 cfu
  Interventions: Biological: BCG TICE strain

INTERVENTIONS:
Biological: BCG TICE strain — All doses: Tice Bacillus Calmette-Guerin (BCG) will be administered as a single 0.1 ml ID injection over the deltoid muscle of the preferred arm. Groups 1 - 4 will receive one dose of Tice BCG intradermally at 2x10^6 cfu, 4x10^6 cfu, 8x10^6 cfu and 16x10^6 cfu, respectively.

SUMMARY:
This is a Phase I open-label, dose escalation trial to evaluate the use of Tice® BCG as a challenge for future assessment of in vivo TB immunity. Subjects will be recruited from the target population reflecting the community at 2 VTEU sites. Enrollment will occur over 14 months. Subjects who provide informed consent will be screened, and up to 120 eligible, HIV and TB uninfected subjects, 18-45 years, inclusive, will be enrolled for study interventions and sequentially assigned to 1 of 4 dose groups. Doses of Tice BCG from 2 to 16x10^6 cfu will be delivered ID in a dose escalation format to 4 groups of 30 subjects per dose group. Primary Objectives: 1) Evaluate the safety of different doses of ID Tice BCG for use as a human challenge model for TB infection. 2) Examine shedding from ID challenge sites after administration of different doses of Tice BCG in TB naive healthy subjects. 3) Evaluate the reproducibility of BCG shedding over time with both quantitative PCR and culture.

DETAILED DESCRIPTION:
This is a Phase I open-label, dose escalation trial to evaluate the use of Tice® BCG as a challenge for future assessment of in vivo TB immunity. Subjects will be recruited from the target population reflecting the community at large at 2 VTEU sites. It is anticipated that enrollment will occur over a 14-month period. Subjects who provide informed consent will be considered for eligibility (screened), and up to 120 eligible, willing, healthy, HIV and TB uninfected subjects aged 18 to 45 years, inclusive, will be enrolled for study interventions and sequentially assigned to 1 of 4 dose groups. Dose titrations of Tice® BCG from 2x10^6 cfu to 16x10^6 cfu will be delivered intradermally in a dose escalation format to 4 groups of 30 subjects per dose group. In the first dose group, subjects will be immunized intradermally with a single dose of 2x10^6 cfu Tice® BCG. The Tice® BCG doses will be increased sequentially from 2x10^6 cfu to 4x10^6 cfu to 8x10^6 cfu to a maximum dose of 16x10^6 cfu following assessment of safety and reactogenicity data from previous dose groups and sentinel subjects. Following administration of Tice® BCG, intradermal (ID) site reactions will be assessed for at least 30 minutes as well as by memory aid on a daily basis throughout the first 15 days. Subjects will also return to the clinic on Days 22, 25, 29, 32, 36, 39, 43, 46, 50, 53, and 57 to evaluate the ID challenge site, assess for lymphadenopathy if indicated based on review of interim medical history and clinical assessment, and review AEs/SAEs, concomitant medications and health status, and collect and dispose of returned biohazard materials. A final clinic visit will be performed at approximately 3 months (Day 99) following administration of Tice® BCG to evaluate the ID challenge site, assess for lymphadenopathy if indicated based on review of interim medical history and clinical assessment, and review SAEs and health status. At approximately 6 months (Day 181) following administration of Tice® BCG a telephone call will be performed to query for any SAEs that may have occurred since the last visit. Based on this information, subjects may be asked to return to the clinic to be evaluated. The duration of the study for each subject will be up to approximately 7 to 8 months. Primary Objectives: 1) Evaluate the safety of different doses of intradermal Tice® BCG for use as a human challenge model for Mycobacterium tuberculosis infection. 2) Examine BCG shedding from intradermal challenge sites after administration of different doses of Tice® BCG in TB naive healthy subjects. 3) Evaluate the reproducibility of BCG shedding over time with both quantitative PCR and culture techniques. Secondary objectives: 1) Determine a tolerable dose of intradermal Tice® BCG that will induce optimal reproducibility of BCG shedding. 2) Determine the method of mycobacterial quantitation that will result in the least variable results. 3) Characterize the magnitude and kinetics of BCG shedding after intradermal Tice® BCG administration at 4 different doses. Parent protocol to sub-study 12-0096.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria for Study Entry:

* Provide written informed consent prior to initiation of any study procedures.
* Are males or non-pregnant females between the ages of 18 and 45 years, inclusive.
* Women of childbearing potential* in sexual relationships with men must use an acceptable method of preventing conception** from 30 days prior to 3 months after Tice® BCG administration.

  *Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal).

  **Includes, but is not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject receiving Tice® BCG, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
* For women of childbearing potential, negative serum pregnancy test at screening and negative urine pregnancy test within 24 hours prior to enrollment and Tice® BCG administration.
* Are in good health, as judged by the investigator and determined by vital signs (oral temperature, pulse, and blood pressure), medical history and physical examination.
* Have a negative HIV-1 ELISA test.
* Have negative serology tests for hepatitis B surface antigen and hepatitis C virus antibody.
* Have a negative QuantiFERON®-TB Gold test. --Negative is defined as Nil response < 0.8 IU/ml and TB Antigen response minus Nil response < 0.35 IU/mL or TB Antigen response minus Nil response > 0.35 IU/mL and < 25% of Nil response and Mitogen response minus Nil response > 0.5 IU/ml.
* Have a urine dipstick for protein less than 1.
* Have a urine dipstick negative for glucose.
* Ability to understand and complete all study visits as required per protocol and be reachable by telephone.

Exclusion Criteria:

Exclusion Criteria for Study Entry:

-Have a history of suspected, confirmed, treated or have other evidence of active tuberculosis. Symptoms may include recurrent fever, fatigue, night sweats, weight loss, oral ulcers, diarrhea, nausea, vomiting, or bleeding.

-Have any systemic symptoms* within 72 hours before Tice® BCG administration or signs of lymphadenopathy, hepatosplenomegaly, or pulmonary disease by physical examination on day of Tice® BCG administration.

* Includes fever, chills, malaise, fatigue, headache, night sweats, weight loss, nausea, vomiting, bleeding, diarrhea, abdominal pain, rhinorrhea, cough, wheezing, or shortness of breath.

  -Have history of any significant acute or chronic medical conditions* or need for chronic medications that, in the opinion of the investigator, will interfere with immunity or affect safety.
* Includes, but is not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.

  -Have any history of excessive scarring or keloid formation.

  -Have household contact or occupation involving significant contact with someone who is immunocompromised*.
* Includes persons with HIV, AIDs, or active cancer; infants (children < 1 year); pregnant women; or persons who are immunosuppressed for approximately 6 weeks (during the time of active ID lesion drainage).

  -Have a history of epilepsy. (Does not include febrile seizures as a child).
  * Have a pacemaker, prosthetic valve, or implantable cardiac devices.
  * Have a history of bleeding disorder.
  * Have a known allergy to any Tice® BCG components (glycerin, asparagine, citric acid, potassium phosphate, magnesium sulfate, iron ammonium citrate, and lactose).
  * Received blood products or immunoglobulin within 6 months prior to Tice® BCG administration.
  * Received immunotherapy within one year prior to Tice® BCG administration.
  * Received or plan to receive live attenuated vaccines 4 weeks before or after Tice® BCG administration.
  * Received or plan to receive inactivated or killed vaccines 2 weeks before or after Tice® BCG administration.
  * Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period.
* Includes trials that have a study intervention such as a drug, biologic, or device.

  -Received an experimental agent* within 30 days prior to Tice® BCG administration or planned receipt of an experimental agent within 90 days after Tice® BCG administration.
* Includes vaccine, drug, biologic, device, blood product, or medication.

  * Have a history of use of a systemic antibiotic within 14 days prior to Tice® BCG administration or planned use of a systemic antibiotic for 3 months after Tice® BCG administration.
  * Have any medical, psychiatric, occupational, or behavioral problems that make it unlikely for the subject to comply with the protocol as determined by the investigator.
  * Are health care providers at the highest risk of acquiring Mtb infection, such as pulmonologists performing bronchoscopies on TB patients.
  * Are breastfeeding or plan to breastfeed at any given time throughout the study.
  * Have long term use* of high dose oral or parenteral glucocorticoids**, or high-dose inhaled steroids***.
* Defined as taken for 2 weeks or more in total at any time during the past 2 months.

  * High dose defined as prednisone >/= 20 mg total daily dose, or equivalent dose of other glucocorticoids.

    * High dose defined as > 800 mcg/day of beclomethasone dipropionate or equivalent.

If short term corticosteroids are given, then the subject should not receive Tice® BCG or have blood collected for immunogenicity studies within 1 week of steroid administration.

* Have immunosuppression or are taking systemic immunosuppressants as a result of an underlying illness or treatment.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 36 months prior to Tice® BCG administration.
* Any active neoplastic disease.
* Have a pulse rate less than 50 bpm or greater than 100 bpm.
* Have a systolic blood pressure less than 90 mm Hg or greater than 140 mm Hg.
* Have a diastolic blood pressure less than 50 mm Hg or greater than 90 mmHg.
* Have a WBC less than 4.0x10^3/UL or greater than 10.5x10^3/UL.
* Have hemoglobin less than 11.5x10^3/UL (female) or less than 12.5x10^3/UL (male).
* Have a platelet count less than 140x10^3/UL.
* Have a creatinine greater than 1.30 mg/dL.
* Have an ALT (SGPT) greater than 40 IU/L (female) or greater than 55 IU/L (male).
* Have known HIV, Hepatitis B, or Hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Have had a positive PPD skin test in the past or received BCG vaccine (BCG vaccination history will be determined by self-report, country of birth, and/or evidence of BCG scar).
* Have a BMI >35.
* PPD skin test within 2 months prior to Tice® BCG administration or planned receipt during the study other than from participation in this study.
* Oral temperature >/= 100.4°F (>/= 38.0°C) or other symptoms of an acute illness within 3 days before Tice® BCG administration. (Subject may be rescheduled).
* Any medical disease or condition that, in the opinion of the investigator, is a contraindication to study participation*.

  * Includes medical disease or condition that would place the subject at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or their successful completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Serious adverse events related to Tice® BCG administration | Day 1 to Day 181
Summary of distribution, in terms of its precision, of BCG shedding from intradermal challenge sites using subjects' peak shedding, as detected by each of 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). | Following Tice® BCG administration biweekly to Week 6
Summary of distribution, terms of its central tendency (mean or GM), of BCG shedding from intradermal challenge sites at 3 time points, as detected by each of 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). | Following Tice® BCG administration biweekly to Week 6
The number of subjects experiencing Grade 3 (severe) clinical safety laboratory adverse events | Day 1 to Day 181
The number of subjects experiencing Grade 3 (severe) injection site reactions following Tice® BCG administration. | Day 1 to Day 15
The number of subjects experiencing Grade 3 (severe) solicited systemic reactions following Tice® BCG administration | Day 1 to Day 15
The number of subjects in groups 3 and 4 experiencing Grade 3 (severe) injection site reactions. | Between Days 16 and 99 following Tice® BCG administration
The number of subjects spontaneously reporting Grade 3 (severe) adverse events related to Tice® BCG administration following Tice® BCG administration. | Day 1 to Day 56

SECONDARY OUTCOMES:
Summary of distribution of the area under the curve for repeated measures of shedding over time from 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). Summarized in terms of its central tendency (mean or GM) | 8 weeks (56 days) following Tice® BCG administration
Summary of distribution of the area under the curve, in terms of its precision, for repeated measures of shedding over time from 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). | 8 weeks (56 days) following Tice® BCG administration
Summary of distribution, in terms of its precision, of BCG shedding from intradermal challenge sites using subjects' peak shedding, as detected by each of 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). | 8 weeks (56 days) following Tice® BCG administration
Summary of distribution, terms of its central tendency (mean or GM), of BCG shedding from intradermal challenge sites at 3 time points, as detected by each of 3 assays (quantitative PCR, quantitative CFU plating and quantitative MGIT BACTEC culture). | 8 weeks (56 days) following Tice® BCG administration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri

REFERENCES:
- [Derived] Blazevic A, Edwards RL, Xia M, Eickhoff CS, Hamzabegovic F, Meza KA, Ning H, Tennant J, Mosby KJ, Ritchie JC, Girmay T, Lai L, McCullough M, Beck A, Kelley C, Edupuganti S, Kabbani S, Buchanan W, Makhene MK, Voronca D, Cherikh S, Goll JB, Rouphael NG, Mulligan MJ, Hoft DF. Phase 1 Open-Label Dose Escalation Trial for the Development of a Human Bacillus Calmette-Guerin Challenge Model for Assessment of Tuberculosis Immunity In Vivo. J Infect Dis. 2024 May 15;229(5):1498-1508. doi: 10.1093/infdis/jiad441. PMID 38019956